CLINICAL TRIAL: NCT02434432
Title: Music Therapy as a Method of Non-Pharmacological Pain Management in the NICU Setting
Brief Title: Music Therapy for Pain Management in the NICU Setting
Acronym: MTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NUR.LB.02
Record Dates: First submitted 2015-04-20; First posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- condition 1 (Experimental): Infants in this arm will receive their mother's choice of music recorded on an Mp player and delivered via headphones.
  Interventions: Behavioral: music therapy selected by mothers
- condition 2 (Active Comparator): Infants in this arm wil receive a recorded Lullaby music delivered to the infant via headphones.
  Interventions: Behavioral: Music therapy recorded lullaby
- Condition 3 (No Intervention): Infants in this arm will have the headphones applied but no music played.

INTERVENTIONS:
Behavioral: music therapy selected by mothers — mothers' choice of music
  Other Names: condition 1
  Arms: condition 1
Behavioral: Music therapy recorded lullaby — recorded lullaby
  Other Names: condition 2
  Arms: condition 2

SUMMARY:
Background: Music therapy has been recommended as an adjuvant therapy for both preterm infants and mothers throughout their stay in the Neonatal Intensive Care Unit (NICU), and has been shown to have some beneficial effects, although conclusive evidence remains lacking.

Objectives: To study the usefulness of two forms of music, as well as no music, on pain and physiological and behavioral parameters of preterm infants during a heel stick procedure for obtaining blood in the Neonatal Intensive Care Unit (NICU).

Hypotheses: Infants hearing music chosen by their mothers will have less pain and optimal behavioral and physiologic responses as compared to infants who hear the lullaby or no music.

Methods: An analytical observational study with a randomized cross-over design will be utilized.

Inclusion will be stable infants born between 28 to 36 weeks of gestation, with normal hearing. Neonatal Physiologic responses [heart rate (HR), oxygen saturation, (02 sat) and respiratory rate(RR)] and Behavioral States will be recorded before and after the heel stick procedure. Maternal age, education, and pregnancy complications will be also be documented. Pain responses will be recorded using the Neonatal Pain, Agitation and Sedation Scale (NPASS).

Ethical considerations: The study imposes minimal risk on infants. One potential risk is that the infant may become agitated while listening to music, especially if it is time for feeding. Based on previous research, infants tend to calm down while listening to music. However, in the infants who may be hungry or fussy, music exacerbate their agitation. To prevent this from occurring the investigators will not perform the heel stick close to feeding time and the investigators will be vigilantly timing and monitoring the infant's agitation. Because music has been shown to calm infants and stop them from crying, the benefits outweigh this risk.

The heel stick is performed routinely on infants (often 3-6 times a day). The investigators will not perform any additional heel sticks for this study, but will rather intervene during one of the scheduled heel stick procedures.

DETAILED DESCRIPTION:
Background and Significance of Study In the United States about half a million infants are born prematurely every year, approximately 12.3%% of all births (CDC, 2011). These infants require extensive care and are hospitalized for long periods of time in the Neonatal intensive care unit (NICU). They are exposed to a multitude of stressful and painful events which are linked to negative developmental outcomes. (Badr et al., 2010, Orcesi et al., 2012). To reduce stress in the NICU and allow for optimal neurobehavioral function, a range of therapies have been studied. Music therapy is one intervention that has been suggested as a tool for alleviating stress in the NICU (Keith, Russell & Weaver, 2009). Music therapy has long been documented to reduce stress, fatigue, and pain and to enhancing relaxation. A meta-analysis of 30 clinical trials using MT for infants in the NICU (Standley, 2012) concluded that MT had significant benefits on heart rate, behavior states, oxygen saturation, sucking/feeding ability, and length of stay. However, the efficacy of music on pain, physiologic and behavioral responses of preterm infants has not been fully supported. While a recent meta-analysis focusing on preterm infants noted that music therapy has significant benefits especially if it was live music and used early in the infant's NICU stay, other studies have not supported the beneficial effects of music (Alipour et al., 2013).

The American Music Therapy Association (AMTA) defines music therapy as the clinical and evidence-based use of music interventions to address physical, psychological, emotional, cognitive, and social needs of individuals, in order to promote an overall well-being, to relieve stress and alleviate pain. Physiologically music acts by redirecting one's attention away from pain inducers by distraction, inducing rhythmic breathing, and allowing for the systematic and rhythmic release of body tension. It can also trigger the autonomic nervous system to allow relaxation in muscle tone, brain wave frequency, galvanic skin response, and pupillary reflexes (Kaminski, 1996).

The preterm infant and music The benefits of classical music therapy on preterm infants in the NICU have been documented in a few studies. Outcomes measured include improved physiological and behavioral responses. Physiological conditions assessed include higher oxygen saturation levels, decreased heart rate, decreased incidences of episodes of apneas and bradycardias and lower energy expenditures (Amini et al., 2013; Chou, Wang, Chen & Pai, 2003; Keidar Mandel, Mimouni, & Lubetzky 2010) Enhanced behavioral responses include: increased calm, quiet, and alert behavioral states, decreased crying and fussy states and improved feeding behaviors (Keith, Russell & Weaver 2009; Lowey et al 2013). Increased formula intake, increased weight gain and less days of hospitalization have also been reported (Cevasco & Grant, 2005; Standley et al., 2010).

In terms of the effect of music on pain responses which is the main objective of this study, only four studies have been published to date. One study assessed the physiological. behavioral and pain responses of preterm infants during recovery from heel lance in 14 preterm infants at 29 to 36 weeks post-conceptual age (PCA) who listened to Brahms' lullaby. Results showed a more rapid return to baseline heart rate, enhanced behavioral states and less pain in infants who listened to music (Butt & Kisilevsky, 2000). Bo & Callaghan (2000) compared four different types of interventions (non-nutrative sucking (NNS), music therapy (MT), and combined NNS and MT (NNS + MT), and no intervention on 27 infants. Results showed that all three interventions had a significant effect on HR, oxygen saturation and pain with NNS + MT having the strongest effect. Whipple (2008) randomly assigned 60 infants between the ages of 32 to 37 weeks to one of three treatment groups: pacifier-activated lullaby (PAL), pacifier-only, and no-contact. Pacifier-only infants did not receive music reinforcement for sucking, and no-contact infants were not provided a pacifier or music at any point during the procedure. There were no significant differences in physiologic measures between groups; however, infants in the PAL group had lower stress levels during-the heelstick procedure than the no-contact group or the pacifier only group. To test if enhancing kangaroo mother care (KMC) by adding rocking, singing and sucking is more efficacious than simple KMC for procedural pain in preterm neonates 90 preterm infants the GA of 32-36 weeks were randomly assigned to 2 conditions: KMC with the addition of rocking, singing and sucking or the infant was held in KMC without additional stimulation. The results showed no significant differences in conditions (Johnston et al, 2009). To summarize the 4 studies provide inconclusive evidence to benefits of music therapy on pain responses in preterm infants and more research is warranted. Furthermore, a systematic review of randomized controlled trials by Hartling et al., (2009) concluded that the studies on the efficacy of music on the pain responses of preterm infants were of low quality methodologically and more studies are necessary.

The GAP in Research Studies investigating the impact of exposure to any form of auditory stimulation in infants have been complicated by a large range of decibel levels and mode of delivery. A likely explanation for this is that many studies were conducted before or close to the time the American Academy of Pediatrics Committee on Environmental Health was making recommendations for what is now considered safe sound levels within the NICU (hourly Leq of 50 dB, hourly L10 of 55 dB, and 1-second duration Lmax < 70 dB). Furthermore, studies have used different modes of music or auditory stimuli with lack of standardization. No one study has looked at the efficacy of music chosen by mothers and which she had listed to while pregnant which is likely to be the most soothing for infants

Methods Design: An analytical observational study with a randomized cross-over design will be utilized.

Setting: The NICU at the American University of Beirut Medical Center (AUBMC).

Subjects: To achieve a power of 0.8 at α = 0.05 and one-tailed with a medium effect size of 0.61 and a medium correlation (r = 0.50) among two repeated measures using the F-test, a sample size of 40 infant will suffice. This sample size is based on previous studies which show a significant difference on the pain scores and using the following formula:

N = (Zα + Zβ)2 x 2 σ 2 Mean difference 2

Instruments/outcome measures All outcome measures will be recorded by three nurses trained to a reliability above r = 80 on the NPASS and the Behavioral States and who are blinded to the intervention type.

Physiologic measures: Heart rates, oxygen saturation levels and respiratory rates will recorded every 1 minute, (5 minutes before, during and 5 minutes after the heel stick) by observing the monitor Behavioral states: The infant's state will be given a numerical score as follows: 1, deep sleep; 2, light sleep; 3, drowsy; 4, quiet awake or alert; 5, actively awake and aroused; 6, highly aroused, upset, or crying; and 7, prolonged respiratory pause > 8 seconds (Als et al., 2005) Pain assessment: The N-PASS, or Neonatal Pain, Agitation and Sedation Scale will be used to assess pain which is a valid, clinically reliable, age-appropriate method to continuously and systematically assess pain and stressful behavior states in infants with a gestational age of 23 weeks and above and from 0 to 100 days of life (Hummel, Puchalski, Creech, & Weiss, 2008). At AUBMC's NICU, the N-PASS is being used routinely as a pain and agitation tool by all nurses to assess infants' responses to pain.

The intervention: Music therapy which will include either a lullaby used in earlier research studies or the mothers choice of music which she has listened to while the infant was in utero. Music will be delivered by a portable mp3 player through head phones.

Procedure A within-subject, crossover, repeated design will be used with infants acting as their own controls. Infants will receive either the mother's music for 5 minutes, the classical lullabies for 5 minutes or no music before the heel stick procedure which is regularly scheduled for all infants in the NICU. After the heel stick 5 minutes of music will be provided. Noise levels will be assessed continuously 10 cm from the infant's ear with a sound analyzer and a decibel scale filter (407790 Octave Band Sound Analyzer, type 2 Integrating Sound Level Meter and Decibel-A Scale Filter, respectively; Extech Instruments, Melrose, MA, USA). Infants' physiological and behavioral states will be assessed and recorded before and after the heel stick and pain assessment will be done after the heel stick.

Statistical analysis Statistical analysis will be performed using the SPSS for Windows version 22.0 (SPSS Inc., Chicago, IL). Comparisons between interventions will be made using repeated measures analysis of variance (RANOVA), when appropriate for distribution normality and post hoc analysis with Bonferroni adjustment Categorical data were analyzed using the chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Infants will be included if they meet the following criteria: between 28 to 36 weeks gestational age, stable condition, not requiring any respiratory support, in an isolette or open crib, are at least one week post natal age and if their mothers have listened to music while pregnant.

Exclusion Criteria:

* Infant will be excluded if they are intubated and on a ventilator or high frequency ventilation, if they have a congenital anomaly that mainly affects hearing, such as craniofacial anomalies; and if they have brain anomalies associated with neurological disorders such as: grade 3-4 intraventricular hemorrhage and periventricular leukomalacia.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
pain responses of preterm infants assessed on the NPASS | During a heelstick procedure 5 minutes after the music conditions 1 & 2 or the control

SECONDARY OUTCOMES:
Physiologic resposnes | 5 minutes before, during and five minutes after the heelstick
  Physiologic responses: Heart rate, Respiratory rate and Oxygen saturations recorded 5 munites before, during, and 5 minutes after the heelstick.
Behavioral responses | Recorded at 5 minutes before during and five minutes after the heelstick
  Behavioral responses recorded using the Brazelton behavioral scale; 5 minutes before during and five minutes after the heelstick

CONTACTS AND LOCATIONS:
Locations (1):
- American University Medical Center (AUBMC), Beirut, Lebanon

REFERENCES:
- [Background] Orcesi S, Olivieri I, Longo S, Perotti G, La Piana R, Tinelli C, Spinillo A, Balottin U, Stronati M. Neurodevelopmental outcome of preterm very low birth weight infants born from 2005 to 2007. Eur J Paediatr Neurol. 2012 Nov;16(6):716-23. doi: 10.1016/j.ejpn.2012.05.006. Epub 2012 Jun 17. PMID 22709626
- [Background] Keith DR, Russell K, Weaver BS. The effects of music listening on inconsolable crying in premature infants. J Music Ther. 2009 Fall;46(3):191-203. doi: 10.1093/jmt/46.3.191. PMID 19757875
- [Background] Standley J. Music therapy research in the NICU: an updated meta-analysis. Neonatal Netw. 2012 Sep-Oct;31(5):311-6. doi: 10.1891/0730-0832.31.5.311. PMID 22908052
- [Background] Alipour Z, Eskandari N, Ahmari Tehran H, Eshagh Hossaini SK, Sangi S. Effects of music on physiological and behavioral responses of premature infants: a randomized controlled trial. Complement Ther Clin Pract. 2013 Aug;19(3):128-32. doi: 10.1016/j.ctcp.2013.02.007. Epub 2013 May 9. PMID 23890458
- [Background] Badr LK, Abdallah B, Hawari M, Sidani S, Kassar M, Nakad P, Breidi J. Determinants of premature infant pain responses to heel sticks. Pediatr Nurs. 2010 May-Jun;36(3):129-36. PMID 20687304
- [Background] Kaminski J, Hall W. The effect of soothing music on neonatal behavioral states in the hospital newborn nursery. Neonatal Netw. 1996 Feb;15(1):45-54. PMID 8700082
- [Background] Chen LC, Wu YC, Hsieh WS, Hsu CH, Leng CH, Chen WJ, Chiu NC, Lee WT, Yang MC, Fang LJ, Hsu HC, Jeng SF. The effect of in-hospital developmental care on neonatal morbidity, growth and development of preterm Taiwanese infants: a randomized controlled trial. Early Hum Dev. 2013 May;89(5):301-6. doi: 10.1016/j.earlhumdev.2012.10.008. Epub 2012 Nov 17. PMID 23168303
- [Background] Chou LL, Wang RH, Chen SJ, Pai L. Effects of music therapy on oxygen saturation in premature infants receiving endotracheal suctioning. J Nurs Res. 2003 Sep;11(3):209-16. doi: 10.1097/01.jnr.0000347637.02971.ec. PMID 14579198
- [Background] Whipple J. The effect of music-reinforced nonnutritive sucking on state of preterm, low birthweight infants experiencing heelstick. J Music Ther. 2008 Fall;45(3):227-72. doi: 10.1093/jmt/45.3.227. PMID 18959451
- [Background] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Background] Cevasco AM, Grant RE. Effects of the pacifier activated lullaby on weight gain of premature infants. J Music Ther. 2005 Summer;42(2):123-39. doi: 10.1093/jmt/42.2.123. PMID 15913390
- [Background] Yildiz A, Arikan D. The effects of giving pacifiers to premature infants and making them listen to lullabies on their transition period for total oral feeding and sucking success. J Clin Nurs. 2012 Mar;21(5-6):644-56. doi: 10.1111/j.1365-2702.2010.03634.x. Epub 2011 Jun 13. PMID 21668549
- [Background] Standley JM, Cassidy J, Grant R, Cevasco A, Szuch C, Nguyen J, Walworth D, Procelli D, Jarred J, Adams K. The effect of music reinforcement for non-nutritive sucking on nipple feeding of premature infants. Pediatr Nurs. 2010 May-Jun;36(3):138-45. PMID 20687305
- [Background] Bo LK, Callaghan P. Soothing pain-elicited distress in Chinese neonates. Pediatrics. 2000 Apr;105(4):E49. doi: 10.1542/peds.105.4.e49. PMID 10742370
- [Background] Butt ML, Kisilevsky BS. Music modulates behaviour of premature infants following heel lance. Can J Nurs Res. 2000 Mar;31(4):17-39. PMID 11189668
- [Background] Johnston CC, Filion F, Campbell-Yeo M, Goulet C, Bell L, McNaughton K, Byron J. Enhanced kangaroo mother care for heel lance in preterm neonates: a crossover trial. J Perinatol. 2009 Jan;29(1):51-6. doi: 10.1038/jp.2008.113. Epub 2008 Sep 4. PMID 18769382
- [Background] Hartling L, Shaik MS, Tjosvold L, Leicht R, Liang Y, Kumar M. Music for medical indications in the neonatal period: a systematic review of randomised controlled trials. Arch Dis Child Fetal Neonatal Ed. 2009 Sep;94(5):F349-54. doi: 10.1136/adc.2008.148411. Epub 2009 May 28. PMID 19477913
- [Background] Hummel P, Puchalski M, Creech SD, Weiss MG. Clinical reliability and validity of the N-PASS: neonatal pain, agitation and sedation scale with prolonged pain. J Perinatol. 2008 Jan;28(1):55-60. doi: 10.1038/sj.jp.7211861. Epub 2007 Oct 25. PMID 18165830
- [Background] Als H, Lawhon G, Brown E, Gibes R, Duffy FH, McAnulty G, Blickman JG. Individualized behavioral and environmental care for the very low birth weight preterm infant at high risk for bronchopulmonary dysplasia: neonatal intensive care unit and developmental outcome. Pediatrics. 1986 Dec;78(6):1123-32. PMID 3786036